CLINICAL TRIAL: NCT04894084
Title: Investigation of a Supporting Ostomy Product Intended for Leakage Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CP321
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-08

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Intervention Model Description: Single arm, open label study. Subjects are allocated to use test product for 3 weeks. Subjects will complete questionnaires at baseline (V1) and again after 3 weeks use of test product (V2). Comparative tests included: Baseline vs. follow-up measures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test product (Experimental): Subjects are requested to use the test device (supporting product) beneath their ostomy baseplate. Subjects may change their appliance as they wish, either they may change due to a notification from the app and/or follow their change routine.
  Interventions: Device: CP321

INTERVENTIONS:
Device: CP321 — The primary objective is to evaluate the system performance of the test product. This is done by asking subjects to answer questions throughout the study

SUMMARY:
People with intestinal stomas (especially an ileostomy) can have, despite development of better ostomy products, problems with leakage which influence their quality of life negatively.

To overcome this, Coloplast has developed a new supporting ostomy product, which has an adhesive sensor layer that should be place underneath the baseplate normally used by the subject.

Single arm design. Open-labelled Study duration: 21 days + 3 days.

DETAILED DESCRIPTION:
Test product is a Digital Leakage Notification System. It consist of a sensor layer (worn beneath the baseplate), a transmitter attached to the sensor layer, a charger for charging of transmitter and an app, to be installed on a smartphone, which notifies the user of the status of their baseplate such as everything looks okay or there is a possible leakage.

Subjects are asked to use test product for 21 days. n=15 were using a phone with Android operating system and n=10 a phone with iOS operating system.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had a stoma for more than three months
4. Have intact skin on the area used in the evaluation meaning no broken skin and only minor discoloration of the skin (assessed by investigator)
5. Be able to use one of the five sensor layer sizes (i.e. Ø40, Ø50, Ø60, Ø70, Ø80 mm)
6. Ileo- or colostomists with liquid output (Bristol scale type 6-7).
7. Currently using a Coloplast product (1pc/2pc Flat/Convex/Concave) from e.g Assura/SenSura/SenSura Mio
8. Have self-reported problems with leakage* (three times within 14 days)
9. Have worry of leakage 'to some, high or very high degree'
10. Is familiar with the use of a smartphone *Leakage: Leakage is defined as output from the stoma on the backside of the baseplate (underneath the baseplate)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Participating in other interventional clinical investigations or have previously participated in this investigation. Exception: Participation in other Coloplast sponsored clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this protocol.
5. Known sensitivity towards test product
6. Known sensitivity towards acrylate
7. Is using/have a pacemaker
8. Is using ostomy paste or ostomy powder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren Meisner, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brady RR, Fellows J, Meisner S, Olsen JK, Vestergaard M, Ajslev TA. A pilot study of a digital ostomy leakage notification system: impact on worry and quality of life. Br J Nurs. 2023 Mar 23;32(6):S4-S12. doi: 10.12968/bjon.2023.32.6.S4. PMID 36952372

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Arm, Intention to Treat: All subjects enrolled into the study (n=25) who have at least one measure on any of the outcomes measured.
  Single arm, open-label investigation with subjects assigned to use test product for 21±3 days.
  Due to technical reasons, data from the questionnaire at V2 for two subjects could not be retrieved from the phones and therefore have been omitted from statistical analyses. Data from the two subjects provided at V1 were included, whenever possible. Therefore, the total number of subjects in the statistical analyses at V1 was n=25, while at V2 the number was n=23.
Period: Overall Study
Arm/Group | Test Arm, Intention to Treat
Started (Enrollment started April 29th 2021) | 25
Completed (Study completed (Last patient out July 14th 2021)) | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Test Arm, Intention to Treat: All subjects enrolled into the study (n=25) who have at least one measure on any of the outcomes measured.
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 56 [36 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All 25 subjects were recruited in Denmark
  Participants
    Denmark | 25
Type of stoma [Count of Participants; unit: Participants]
  Ileostomy | 15
  Colostomy | 10

OUTCOME MEASURES:

1. Primary Outcome: System Performance Accuracy of Pictures
Description: The primary endpoint is system performance accuracy:
  * True Negative: No leakage observed on picture and no leakage detected by system
  * True Positive: Leakage observed in picture and leakage detected by system
  * False Negative: Leakage observed in picture, but no leakage detected by system
  * False Positive: No leakage observed in picture, but leakage detected by system
Time Frame: 21 days
Measure: Count of Units; unit: Pictures
Units Other Than Participants: Pictures
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 25
Number analyzed (Pictures) | 317
Pictures
  True positive | 122
  True negative | 126
  False positive | 24
  False negative | 45

2. Secondary Outcome: Frequency of Leakage Onto Clothes Before and After Use of Test Product
Description: Subjects are asked to recall numbers of leakage events outside baseplate (and/or onto clothes) the past 3 weeks (at baseline and follow-up). Subjects shall give a specific frequency.
Time Frame: At V1 (baseline) and V2 (follow-up, Day 21)
Measure: Least Squares Mean (95% Confidence Interval); unit: Leakage episodes onto clothes
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 25
Leakage episodes onto clothes
  V1 | 2.84 [1.69 to 4.76]
  V2 | 0.51 [0.19 to 1.36]
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Superiority; p < 0.001, Poisson loglinear model; Risk Ratio (RR) = 0.18, 95% CI 2-sided [0.07 to 0.49]

3. Secondary Outcome: Experience of Leakage Onto Clothes Compared to Only Using Usual Product
Description: Subject own interpretation, Q: to which degree have you experienced leakage onto your clothes with test product?" (5-point scale: very low degree/not at all, low degree, some degree, high degree, very high degree).
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Very high degree | 0
  High degree | 0
  Some degree | 2
  Low degree | 3
  Very low degree / Not at all | 18
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; For secondary endpoints where the possible answer is Yes or No, the proportion of subjects answering "Yes" was calculated. By use of an exact test in the binomial distribution a 95% confidence interval was estimated for the proportion. It was tested if the proportion was significantly different from 50% when using a 5% test level. For questions answered on a 5-point scale the answers was grouped in 2 (e.g. "higher" or "much higher" against the rest of the answers); Test type: Other; p < 0.0001, Exact test in the binomial distribution — "Low degree" + "Very low degree / Not at all" were tested against the rest of the answers in this analysis; Exact test in the binomial distribution = 91.3, 95% CI 2-sided [72 to 99]

4. Secondary Outcome: Reliability of Notifications
Description: Subjects are asked to rate, Q: To which degree did you find notifications from the app reliable and trustworthy (5-point scale; very low degree, low degree, some degree, high degree, very high degree)
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Very high degree | 5
  High degree | 7
  Some degree | 6
  Low degree | 3
  Very low degree / Not at all | 2
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; For secondary endpoints an exact test in the binomial distribution a 95% confidence interval was estimated for the proportion. It was tested if the proportion was significantly different from 50% when using a 5% test level. For reliability answered on a 5-point scale the answers some, high, or very high degree was considered acceptable and grouped against answers of 'low or very low' degree of reliability; Test type: Other; p = 0.0106, Exact test in the binomial distribution — "Some degree", "High degree" and "Very high degree" were tested against the rest of the answers in this analysis; Exact test in the binomial distribution = 78.3, 95% CI 2-sided [56 to 93]

5. Secondary Outcome: Ability to Move With Test Product
Description: Q: Compared to your usual product, how was your freedom to move with test product? Much better - better - Same - Worse - Much worse
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Much worse | 0
  Worse | 1
  Same | 16
  Better | 4
  Much better | 2
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; For secondary endpoints an exact test in the binomial distribution a 95% confidence interval was estimated for the proportion. For ability to move with test product it was tested if the proportion evaluating same or better was significantly different from 50% when using a 5% test level. The answers of 'same, better or much better' was grouped against the answers of 'worse or much worse' ability to move; Test type: Other; p < 0.0001, Exact test in the binomial distribution — "Same", "Better" and "Much better" were tested against the rest of the answers in this analysis; Exact test in the binomial distribution = 95.7, 95% CI 2-sided [78 to 100]

6. Secondary Outcome: Subjects Worry of Leakage Before and After Use of Test Product
Description: Q: Think back on the last 3 weeks - to which degree have you worried about leakage? Very high degree - High degree - Some degree - Low degree - Very low degree/Not at all
Time Frame: At V1 (baseline) and V2 (follow-up, Day 21)
Population: Due to technical reasons, data from the questionnaire at V2 for two subjects could not be retrieved from the phones and therefore have been omitted from statistical analyses. Data from the two subjects provided at V1 were included, whenever possible. Therefore, the total number of subjects in the statistical analyses at V1 was n=25, while at V2 the number was n=23.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 25
Participants
  V1: Very high degree | 1
  V1: High degree | 11
  V1: Some degree | 11
  V1: Low degree | 2
  V1: Very low degree / Not at all | 0
  V2: number analyzed (Participants) | 23
  V2: Very high degree | 0
  V2: High degree | 1
  V2: Some degree | 6
  V2: Low degree | 8
  V2: Very low degree / Not at all | 8
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — Users worry of leakage given on a 5-point scale was analyzed by a proportional odds ratio model taken the paired design into consideration to compare the results from V1 and V2; p < 0.001, Proportional odds ratio model

7. Secondary Outcome: Confidence to Avoid Full Leakage With Test Product Compared to Only Using Usual Product
Description: Q: Compared to your usual product, did you feel confident that you could avoid leakage onto clothes? Yes -No
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Yes | 18
  No | 5
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — For secondary endpoints where the possible answer is Yes or No, the proportion of subjects answering "Yes" was calculated. By use of an exact test in the binomial distribution a 95% confidence interval was estimated for the proportion. It was tested if the proportion was significantly different from 50% when using a 5% test level; p = 0.0106, Exact test in the binomial distribution; Exact test in the binomial distribution = 78.3, 95% CI 2-sided [56 to 93]

8. Secondary Outcome: Confidence in Daily Life Compared to Only Using Usual Product
Description: Q: Compared to your usual product, to which degree did the test product give you confidence in daily life? Much higher degree- Higher degree- Same degree - Lower degree- Much lower degree
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Much lower degree | 1
  Lower degree | 2
  Same degree | 5
  Higher degree | 10
  Much higher degree | 5
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — For secondary endpoints where the possible answer is Yes or No, the proportion of subjects answering "Yes" was calculated. By use of an exact test in the binomial distribution a 95% confidence interval was estimated for the proportion. It was tested if the proportion was significantly different from 50% when using a 5% test level. For questions answered on a 5-point scale the answers was grouped in 2 (e.g. "higher" or "much higher" against the rest of the answers); p = 0.21, Exact test in the binomial distribution — "Higher degree" and "Much higher degree" were tested against the rest of the answers in this analysis; Exact test in the binomial distribution = 65.2, 95% CI 2-sided [43 to 84]

9. Secondary Outcome: Feeling of Control With Test Product Compared to Only Using Usual Product
Description: Q: Compared to your usual product, did test product give you a feeling of leakage control? Yes, higher leakage control No, lower leakage control
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Yes, higher leakage control | 18
  No, lower leakage control | 5
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0106, Exact test in the binomial distribution; Exact test in the binomial distribution = 78.3, 95% CI 2-sided [56 to 93]

10. Secondary Outcome: Control of Leakage Progression With Test Product Compared to Only Using Usual Product
Description: Q: Compared to your usual product, did the test product give you a feeling of control of leakage progression? Yes, higher control of leakage progression No, lower control of leakage progression
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Yes, higher control of leakage progression | 16
  No, lower control of leakage progression | 7
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.093, Exact test in the binomial distribution; Exact test in the binomial distribution = 69.6, 95% CI 2-sided [47 to 87]

11. Secondary Outcome: Feeling of Security With Test Product Compared to Only Using Usual Product
Description: Q: Compared to your usual product, did you feel more or less secure with test product?
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  I felt less secure | 1
  I felt more secure | 22
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — By use of an exact test in the binomial distribution a 95% confidence interval was estimated for the proportion. It was tested if the proportion with a positive response was significantly different from 50% when using a 5% test level; p < 0.0001, Exact test in the binomial distribution; Exact test in the binomial distribution = 95.7, 95% CI 2-sided [78 to 100]

12. Secondary Outcome: Evaluation of Confidence to Increase Social Activities With Test Product Compared to Only Using Usual Product
Description: Q: Compared with your usual product, did the test product affect your confidence to engage in social activities such as seeing friends, and do physical activities? I felt more confident - I felt less confident
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  I felt less confident | 2
  I felt more confident | 21
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — By use of an exact test in the binomial distribution a 95% confidence interval was estimated for the proportion. It was tested if the proportion answering I felt more confident was significantly different from 50% when using a 5% test level; p < 0.0001, Exact test in the binomial distribution; Exact test in the binomial distribution = 91.3, 95% CI 2-sided [72 to 99]

13. Secondary Outcome: Evaluation of Sleep With Test Product Compared to Only Using Usual Product
Description: Q: Compared with your usual product, did the test product affect your sleep? Yes, to the better Yes, to the worse No, the same
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Yes, to the better | 8
  Yes, to the worse | 0
  No, the same | 15
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.21, Exact test in the binomial distribution — "Yes, to the better" was tested against the rest of the answers in this analysis; Exact test in the binomial distribution = 34.8, 95% CI 2-sided [16 to 57]

14. Secondary Outcome: Confidence at Night With Test Product Compared to Only Using Usual Product
Description: Compared with your usual product, to which degree did the test product give you confidence at night? Much higher - Higher - Same - Lower - Much lower
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Much lower degree | 0
  Lower degree | 1
  Same degree | 11
  Higher degree | 7
  Much higher degree | 4
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 1.00, Exact test in the binomial distribution — "Higher degree" and "Much higher degree" were tested against the rest of the answers in this analysis; Exact test in the binomial distribution = 47.8, 95% CI 2-sided [27 to 69]

15. Secondary Outcome: Evaluation of Users' Preference
Description: Q: Which product solution do you prefer? Own product - Own product with test product
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Own product | 10
  Own product with test product | 13
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.678, Exact test in the binomial distribution; Exact test in the binomial distribution = 56.5, 95% CI 2-sided [34 to 77]

16. Secondary Outcome: Reason for Preference
Description: Q: What is your reason for preference? (Please tick all that apply)
  * Body fit
  * Ability to bend and stretch
  * Feeling of security
  * Feeling of confidence
  * Less fear of leakage onto clothes
  * Discreet to wear
  * Discreetness in leakage control
  * Better sleep
  * Less embarrassment
  * Other
Time Frame: V2 (follow-up, Day 21)
Population: The 13 subjects with a preference for test product were asked for the reason(s) for this preference and the the 10 subjects with a preference for own product were asked for the reason(s) for this preference.
Measure: Number; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Preference for test product : Body fit: number analyzed (Participants) | 13
  Preference for test product : Body fit | 2
  Preference for test product : Ability to bend and stretch: number analyzed (Participants) | 13
  Preference for test product : Ability to bend and stretch | 1
  Preference for test product : Feeling of security: number analyzed (Participants) | 13
  Preference for test product : Feeling of security | 10
  Preference for test product : Feeling of confidence: number analyzed (Participants) | 13
  Preference for test product : Feeling of confidence | 2
  Preference for test product : Less fear of leakage onto clothes: number analyzed (Participants) | 13
  Preference for test product : Less fear of leakage onto clothes | 9
  Preference for test product : Discreet to wear: number analyzed (Participants) | 13
  Preference for test product : Discreet to wear | 2
  Preference for test product : Discreetness in leakage control: number analyzed (Participants) | 13
  Preference for test product : Discreetness in leakage control | 10
  Preference for test product : Better sleep: number analyzed (Participants) | 13
  Preference for test product : Better sleep | 5
  Preference for test product : Less embarrassment: number analyzed (Participants) | 13
  Preference for test product : Less embarrassment | 1
  Preference for test product : Other: number analyzed (Participants) | 13
  Preference for test product : Other | 0
  Preference for own product : Body fit: number analyzed (Participants) | 10
  Preference for own product : Body fit | 5
  Preference for own product : Ability to bend and stretch: number analyzed (Participants) | 10
  Preference for own product : Ability to bend and stretch | 3
  Preference for own product : Feeling of security: number analyzed (Participants) | 10
  Preference for own product : Feeling of security | 3
  Preference for own product : Feeling of confidence: number analyzed (Participants) | 10
  Preference for own product : Feeling of confidence | 0
  Preference for own product : Less fear of leakage onto clothes: number analyzed (Participants) | 10
  Preference for own product : Less fear of leakage onto clothes | 1
  Preference for own product : Discreet to wear: number analyzed (Participants) | 10
  Preference for own product : Discreet to wear | 3
  Preference for own product : Discreetness in leakage control: number analyzed (Participants) | 10
  Preference for own product : Discreetness in leakage control | 4
  Preference for own product : Better sleep: number analyzed (Participants) | 10
  Preference for own product : Better sleep | 0
  Preference for own product : Less embarrassment: number analyzed (Participants) | 10
  Preference for own product : Less embarrassment | 0
  Preference for own product : Other: number analyzed (Participants) | 10
  Preference for own product : Other | 1

17. Secondary Outcome: Evaluation of Users' Peace of Mind With Test Product
Description: Q: To which degree did the test product give you peace of mind? Very high degree- High degree- Low degree- Very low degree
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Very high degree | 6
  High degree | 10
  Low degree | 5
  Very low degree | 2
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0931, Exact test in the binomial distribution — "High degree" and "Very high degree" were tested against the rest of the answers in this analysis; Exact test in the binomial distribution = 69.6, 95% CI 2-sided [47 to 87]

18. Secondary Outcome: To Evaluate Users' Assessment of QoL With Test Product Compared to Usual Product
Description: Overall, do you think the test product can improve your feeling of control and confidence to avoid leakage onto clothes and therefore improve your quality of life? Yes - No
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  No | 3
  Yes | 20
Statistical Analysis 1: Comparison: Test Arm, Intention to Treat; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.0005, Exact test in the binomial distribution; Exact test in the binomial distribution = 87.0, 95% CI 2-sided [66 to 97]

19. Secondary Outcome: Adhesive Residue to Skin
Description: To which degree did you experience adhesive residue to the skin in the area around the transmitter? Very low degree/Not at all - Low degree - Some degree - High degree -Very high degree
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Very low degree/Not at all | 6
  Low degree | 7
  Some degree | 7
  High degree | 2
  Very high degree | 1

20. Secondary Outcome: Adhesive Residue to Transmitter
Description: To which degree did you experience adhesive residue on the backside of the transmitter? Very low degree/Not at all - Low degree - Some degree - High degree -Very high degree
Time Frame: V2 (follow-up, Day 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm, Intention to Treat
Number analyzed (Participants) | 23
Participants
  Very low degree/Not at all | 9
  Low degree | 5
  Some degree | 9
  High degree | 0
  Very high degree | 0

ADVERSE EVENTS:
Time Frame: 21 days
Description: During Visit 2, potential (S)AE's was captured by the Principal Investigator, or delegate.
Arm/Group | Test Product
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=25)
Skin redness and irritation (Skin and subcutaneous tissue disorders) | 2 (2) — Red and irritated skin in the area where the leg of the sensorplate has been placed. Possibly or probably related to the device. Intensity: Mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT04894084/Prot_SAP_001.pdf